CLINICAL TRIAL: NCT05733104
Title: Prospective Observational Post Marketing Surveillance Study to Observe Safety and Effectiveness of Zavicefta IV
Brief Title: A Study to Learn About the Study Medicine Zavicefta After it is Released Into the Markets in Korea
Status: Recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C3591027
Record Dates: First submitted 2022-12-12; First posted 2023-02-17 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Complicated Intra-abdominal Infection; Complicated Urinary Tract Infection; Hospital-acquired Pneumonia
Keywords: Ceftazidime; Avibactam; safety; efficacy
MeSH Terms: conditions — Healthcare-Associated Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to learn about the safety and effectiveness of Zavicefta once released into the markets in Korea. This study is to learn about Zavicefta in patients with difficult types of infections in the abdomen, urinary tract and pneumonia which could have come from hospitalizations.

This study was required by the Ministry of Food and Drug Safety (MFDS) of Korea's regulations.

DETAILED DESCRIPTION:
The objective of this study is to determine any problems or questions associated with Zavicefta after marketing, with regard to the following clauses under conditions of general clinical practice, in compliance with the regulation "Re-examination Guideline of New Drugs".

1. Serious adverse event/adverse drug reaction
2. Unexpected adverse event/adverse drug reaction that have not been reflected in the approved drug label.
3. Known adverse drug reaction
4. Non-serious adverse drug reaction
5. Other safety and effectiveness information As required for any new medication approved by Ministry of Food and Drug Safety (MFDS), information on safety and effectiveness of new medication should be researched on certain number of subjects taking the drug in the setting of routine practice during the initial 6 years after the approval of new drug. This reserach shall begin after approval of marketing in Korea by MFDS.

ELIGIBILITY:
1. Adults and paediatric patients aged 3 months and older, who have been administered at least one dose of Zavicefta for the treatment of one of the indications as follows:

   * Complicated intra-abdominal infection (cIAI)
   * Complicated urinary tract infection (cUTI), including pyelonephritis
   * Hospital-acquired pneumonia (HAP), including ventilator associated pneumonia (VAP)
   * Other aerobic Gram-negative organism infection with limited treatment options
2. Adults 19 years of age or older, who have been administered at least one dose of Zavicefta for the treatment of the indication as follows:

   •Bacteremia associated with or suspected to be associated with cIAI, cUTI or HAP including VAP.
3. Patients are treated with Zavicefta for the first time
4. Patients have signed the data privacy statement.

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: At least 600 subjects who are eligible for Zavicefta IV accoding to its product label will be enrolled by continuous registration method and will be researched under routine clinical setting of Korea.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2029-09-28 (Estimated); Study Completion 2029-09-28 (Estimated)

PRIMARY OUTCOMES:
Number of patient reporting an adverse event | From first dose to end of the observation period (at least 28 calendar days following the last dose)
  Safety will be assessed based on adverse events reported for all patients who received at least one dose of Zavicefta and completed safety follow-up.

SECONDARY OUTCOMES:
Clinical response: Number of patient recorded as cure | up to one year
  Clinical response will be evaluated as follows based on subjective assessment by the investigator after the patient has been subjected to the conditions corresponding to each clinical response item or after interviewing the patient at the end of treatment:
  Cure: Complete resolution or significant improvement of signs and symptoms of the index infection, such that no further antibacterial therapy was necessary
  Failure: Death related to the index infection or received treatment with additional antibiotics for ongoing symptoms of index infection
  Indeterminate: study data were not available for evaluation of effectiveness for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3591027